CLINICAL TRIAL: NCT06368219
Title: Propofol or Benzodiazepine Combined With Ketamine for Procedural Sedation in Emergency Setting
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0108161
Record Dates: First submitted 2024-03-29; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Procedural Sedation
Keywords: midazolam; propofol; ketamine; procedural sedation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- midazolam- ketamine combination (Active Comparator): - Group A: 25 patients will receive ketamine (0.5 mg/kg) plus midazolam (0.05 mg/kg
  Interventions: Drug: ketamine- midazolam versus ketamine- propofol
- propofol- ketamine combination (Active Comparator): - Group B: 25 patients will receive ketamine (0.5 mg/kg) plus propofol (0.5 mg/kg)(
  Interventions: Drug: ketamine- midazolam versus ketamine- propofol

INTERVENTIONS:
Drug: ketamine- midazolam versus ketamine- propofol — * Group A: 25 patients will receive ketamine (0.5 mg/kg) plus midazolam (0.05 mg/kg)
  * Group B: 25 patients will receive ketamine (0.5 mg/kg) plus propofol (0.5 mg/kg)

SUMMARY:
This single blinded parallel randomized clinical trial will be conducted on 50 patients presented to Emergency Department of Alexandria Main University Hospital who are indicated for procedural sedation. All patients included in the study will be allocated randomly using computer software with concealment of randomization in to two groups:

* Group A: 25 patients will receive ketamine (0.5 mg/kg) plus midazolam (0.05 mg/kg)
* Group B: 25 patients will receive ketamine (0.5 mg/kg) plus propofol (0.5 mg/kg) Additional ketamine (0.25 mg/kg) will be administered in case of inadequate sedation in both groups.

the two groups will be compared as regard incidence of complications World Society of Intravenous Anesthesia (SIVA) international sedation task force to standardize reporting adverse events

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) requiring procedural sedation and analgesia for painful procedures in ED . The following procedures are indications for PSA:
* Cardioversion
* Reduction of fracture or joint dislocation
* Procedures as central venous catheter (CVC) and chest tube insertion or wound management

Exclusion Criteria:

* Patients with anticipated difficult airway.
* Post cardiac arrest patients.
* Contraindication to study drugs.
* Pregnant women.
* Patients > 65 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Induction and recovery time for both combinations | 2 hours
  the induction and recovery time of ketamine/midazolam versus ketamine/propofol combinations used for procedural sedation in an Emergency setting.

SECONDARY OUTCOMES:
incidence and severity of adverse events | 2 hours
  7) Incidence of complications between the two groups using World Society of Intravenous Anesthesia (SIVA) international sedation task force to standardize reporting adverse events

IPD SHARING:
Plan to Share IPD: No